CLINICAL TRIAL: NCT02872454
Title: Psychotherapeutic Text Messaging for Depression Pilot Study
Acronym: TEXT4U
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Paul Pfeiffer, Principal Investigator, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HUM00090058
Record Dates: First submitted 2015-09-01; First posted 2016-08-19 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Major Depression
Keywords: Major Depression; Text Messaging; Guided Self-Help
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Text Messaging (Experimental)
  Interventions: Behavioral: Text Messaging

INTERVENTIONS:
Behavioral: Text Messaging — Each week, enrolled participants will receive daily text messages from one of three randomly assigned psychotherapeutic modalities-cognitive restructuring, behavioral activation, and techniques based on Acceptance and Commitment Therapy (ACT)-for a total of 12 weeks. The messages were developed, reviewed, and refined by a multidisciplinary team of experienced therapists, including social workers, psychologists, and psychiatrists.

SUMMARY:
Major depression is the leading cause of disability in the United States and is a major contributor to suicide, a leading cause of premature death. The majority of individuals with depression do not receive adequate pharmacologic or psychotherapeutic treatment due to difficulty accessing services or stopping treatment due to side effects, non-response, or the stigma associated with attending mental health clinic visits. Mobile health information technology services, such as text messaging, have the potential to provide effective self-management support for depression to nearly every adult in the US with depression. Guided self-help via text messaging has been shown to be effective for improving a range of health behaviors as well as symptoms of depression. However, previously studied depression text messaging services have not utilized the breadth of psychotherapeutic techniques shown to be effective for depression nor have they attempted to tailor the psychotherapeutic content to the individual in order to improve acceptability and outcomes. Advanced artificial intelligence methods (e.g., reinforcement learning) offers the capability to weed out ineffective messages and to target messages to individuals in order to substantially improve program effectiveness. This pilot study is the first step in towards developing an artificially intelligent text message service for depression.

The specific aims of the study are to: 1) demonstrate the feasibility of recruiting and enrolling participants from the general population of US adults and delivering a text-messaging intervention for depression, 2) determine whether there are differences in the perceived helpfulness of messages derived from different psychotherapeutic treatment modalities, and whether these differences are moderated by participant characteristics (e.g., age, gender, depression symptom severity), 3) determine whether messages derived from different psychotherapeutic treatment modalities or their perceived helpfulness are associated with changes in depression symptoms, and whether these relationships are moderated by participant characteristics.

ELIGIBILITY:
Inclusion Criteria:

* US resident
* Age 18 or older
* PHQ-9 screening score of 10 or more
* Has a personal cellular phone with a text messaging plan that would allow for as many as 200 additional text messages per month, and agreement that the participant would be responsible for any related charges
* Has a valid e-mail address
* Fluent in English

Exclusion Criteria:

* Unable to provide voluntary informed consent for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2015-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Intervention Feasibility | 6 and 12 weeks post-baseline
  Study team's ability to deliver the intervention as a measure of feasibility. Measured by at least 50% of patients who complete the screening questionnaire choosing to enroll in the study, at least 70% of participants completing follow-up measures at 12 weeks, and the study meeting its enrollment goal of 250 patients in 12 months.

SECONDARY OUTCOMES:
Perceived Helpfulness of Messages | baseline and12 weeks post-baseline
  Patient's belief that the program will be helpful as measured by the Credibility/Expectancy Questionnaire and patient's rating of the program at 12 weeks post-baseline as measured by the Study Experience Questionnaire.
Change in Depression Symptoms | 6 and 12 weeks post-baseline
  Patient's current level of depressive symptoms as measured by the Patient Health Questionnaire (PHQ-9).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan Inpatient Psychiatry Unit, Ann Arbor, Michigan, United States